CLINICAL TRIAL: NCT02725632
Title: Sodium Channel Splicing in Obstructive Sleep Apnea (SOCS-OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 411013
Record Dates: First submitted 2016-03-14; First posted 2016-04-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sodium channel; splicing variant; sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): An age-matched control group will be enrolled and consented. A Data Collection Sheet will be used to document data from the subject's medical records including history, physical exam, active medications, laboratory data, polysomnogram, electrocardiogram, echocardiography and cardiac catheterization.
  At the time of enrollment, one blood drawn through peripheral venipuncture will be collected. Another blood drawn will be collected after one month. The blood samples will be processed and analyzed to assess for levels of SCN5A mRNA splicing variants.
- OSA (Active Comparator): Newly diagnosed OSA patients will be enrolled and consented. A Data Collection Sheet will be used to document data from the patient's medical records including history, physical exam, active medications, laboratory data, polysomnogram, electrocardiogram, echocardiography and cardiac catheterization.
  At the time of enrollment, one blood drawn through peripheral venipuncture will be collected. The patients on CPAP treatment will be followed-up for 1 month. Another blood drawn will be collected after one month of CPAP treatment. The blood samples will be processed and analyzed to assess for levels of SCN5A mRNA splicing variants.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — The patients on CPAP treatment will be followed-up for 1 month.
  Arms: OSA

SUMMARY:
This study is designed to test whether SCN5A mRNA processing is altered in OSA patients, which may contribute to their increased arrhythmic risk, and whether processing of SCN5A mRNA is modulated by CPAP treatment.

Specific aims:

1. Compare sodium channel splicing variants in mild, moderate, or severe OSA patients at baseline to at 1 month after CPAP treatment. In addition, the baseline splicing variants of SCN5A in the OSA patients will be compared to an age-matched control group.
2. Hypoxia-associated upstream regulators of SCN5a mRNA splicing, Hypoxia-inducible factor 1-alpha (HIF-1α), RNA Binding Motif Protein 25 (RBM25) and LUC7-Like 3 Pre-MRNA Splicing Factor (LUC7L3), will be examined in OSA patients before and after 1 month of CPAP treatment.

DETAILED DESCRIPTION:
BACKGROUND & SIGNIFICANCE Obstructive sleep apnea (OSA) is a common disease with an estimated prevalence of 3% to 7%. It is characterized by recurrent episodes of partial or complete collapse of the upper airway during sleep, resulting in hypopneas or apneas, respectively. The collapse of upper airway during obstructed events result in intermittent hypoxia, recurrent arousals from sleep, metabolic disturbance and poor quality of life. Cardiac arrhythmias are reportedly more frequent in patients with OSA and increase with the number of apneic episodes and the severity of the associated hypoxemia. Recent data from the Sleep Heart Health Study suggested that those with severe sleep disorders had a 2- to 4-fold-higher risk of nocturnal complex arrhythmias. Even after adjustment for age, sex, BMI, and prevalent coronary artery disease, patients with sleep disorders had increased likelihoods of atrial fibrillation, nonsustained ventricular tachycardia, and complex ventricular ectopy.

Continuous positive airway pressure (CPAP) is the first-line treatment for patients with OSA and acts as a pneumatic splint to the upper airway during sleep and corrects the obstruction, improving daytime sleepiness and quality of life. Observational studies suggest that CPAP treatment reduces the incidence of cardiovascular events in patients with moderate and sever OSA.

Sodium channel is an integral membrane protein that plays a central role in conduction of the cardiac impulse in myocytes and cells of the His-Purkinje system. It is a multimeric complex consisting of an α and an auxiliary β-subunit. The α subunit, SCN5A is sufficient to express a functional channel. However, β subunit co-expression increases the level of channel expression and alters the voltage dependence of inactivation. Mutations of the sodium channel result in type 3 long QT syndrome (LQT3), Brugada syndrome, atrial fibrillation, congenital sick sinus syndrome, multifocal premature ventricular contractions (PVCs), and dilated cardiomyopathy.

Recently, the investigators have discovered abnormal sodium channel messenger RNA (mRNA) processing in congestive heart failure (CHF) that results in reduced sodium channel to a range known to be associated with sudden cardiac death. Three truncated SCN5A mRNA splicing variants were identified (denoted variant B (E28B), variant C (E28C), and variant D (E28D)). Among them, E28C and E28D abundances were increased 14.2 fold and 3.8 fold respectively in CHF patients compared to controls. The full length SCN5A mRNA (E28A) was decreased by 24.7% in patients with CHF compared to control. Moreover, a key transcriptional regulatory molecule in hypoxia, hypoxia-induced factor 1α (HIF-1α), and hypoxia-induced mRNA splicing factors, such as RBM25 and LUC7L3, were elevated in human CHF tissue and mediated in vitro truncation of SCN5A mRNA.

Thus, this study is designed to test whether SCN5A mRNA processing is altered in OSA patients, which may contribute to their increased arrhythmic risk, and whether processing of SCN5A mRNA is modulated by CPAP treatment.

SPECIFIC AIMS

1. Compare sodium channel splicing variants in mild, moderate, or severe OSA patients at baseline to at 1 month after CPAP treatment. In addition, the baseline splicing variants of SCN5A in the OSA patients will be compared to an age-matched control group.
2. Hypoxia-associated upstream regulators of SCN5a mRNA splicing, HIF-1α, RBM25 and LUC7L3, will be examined in OSA patients before and after 1 month of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

OSA Eligibility Criteria:

1. Age greater than 18 years
2. Able to provide informed consent
3. New diagnosis of OSA by polysomnogram
4. Agree with CPAP treatment

Control Eligibility Criteria:

1. Age greater than 18 years
2. Without OSA
3. Able to provide informed consent

Exclusion Criteria:

1. Not able to give informed consent due to psychological incapacity
2. Chronic use of hypnotics for more than 6 weeks
3. Current drug or alcohol addiction
4. Rhythm other than sinus at enrollment
5. Mandatory and biventricular pacing
6. History of heart transplant or left ventricular assist device (LVAD)
7. Active use of intravenous vasodilators, vasopressors or inotropes
8. Hemodialysis or peritoneal dialysis
9. Active infection including bacteremia
10. Acute coronary syndrome (ACS) within 6 weeks
11. Major trauma or surgery within 6 weeks
12. Malignant neoplastic disease on active treatment including chemotherapy and radiation therapy, or life expectancy less than 1 year
13. Collagen vascular disease on active treatment including steroids and other immunomodulating drugs
14. Systemic steroid use within 6 weeks
15. Concomitant use of investigational drug within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The levels of sodium channel splicing variants that are related to the severity of OSA, change from baseline to one month after CPAP treatment. | Four weeks

SECONDARY OUTCOMES:
The levels of potassium channels that are related to the severity of OSA, change from baseline to one month after CPAP treatment. | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Millman, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Brown University, Lifespan, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt SA; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). ACC/AHA 2005 guideline update for the diagnosis and management of chronic heart failure in the adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure). J Am Coll Cardiol. 2005 Sep 20;46(6):e1-82. doi: 10.1016/j.jacc.2005.08.022. No abstract available. PMID 16168273
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Kannel WB, Plehn JF, Cupples LA. Cardiac failure and sudden death in the Framingham Study. Am Heart J. 1988 Apr;115(4):869-75. doi: 10.1016/0002-8703(88)90891-5. PMID 3354416